CLINICAL TRIAL: NCT01985347
Title: The SAD Study - SLEEP, ANXIETY & DEPRESSION Study A Prospective Cohort Study
Acronym: SAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: Lyell McEwin Hospital (Other Government)
Responsible Party: Principal Investigator, Faisal Ameer, Dr, The Queen Elizabeth Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/13/TQEHLMH/14
Record Dates: First submitted 2013-10-28; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Patients With Anxiety and Depression, Who Have; Obstructive Sleep Apnoea; COPD
MeSH Terms: conditions — Depression; Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obstructive Sleep Apnoea (Active Comparator): Patients with newly diagnosed obstructive sleep apnoea and who have anxiety and depression would be given continuous positive airway pressure (CPAP) treatment.
  Interventions: Device: CPAP
- Chronic obstructive pulmonary disease and western population (No Intervention): (For this group no intervention needed).Patients with COPD, who have anxiety and depression & normal population in Western Adelaide who also have anxiety and depression their prevalence would be compare with patients of Obstructive sleep apnoea.

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure( CPAP)
  Arms: Obstructive Sleep Apnoea

SUMMARY:
The prevalence of anxiety and depression in our OSA population is more than in COPD and the general population of North West Adelaide. (principal hypothesis).

CPAP therapy in OSA population produces a positive effect on the anxiety and depression scale.

The Investigators intend to study the prevalence of anxiety and depression in patients with sleep disorders in comparison to patients with COPD and subsequently, to assess whether CPAP has a role in controlling anxiety and depression in depressed and anxious patients with sleep apnoea.

This is a two phase study, in first phase; investigator will assess the prevalence of anxiety and depression, in a population with sleep disorders to check whether it is different to the prevalence in the COPD population. The prevalence of depression in Sleep Disorder population will also be compared with the Adelaide North Western general population, which was reported in The North West Adelaide Health Study. According to this epidemiological survey, which was conducted from 2008 to 2010, the prevalence of depression in Adelaide North Western general population was 20%.During the second phase of the study investigator will evaluate the effect of CPAP on anxiety and depression scores in the depressed and anxious patients with sleep apnoea by comparing the pre and post CPAP anxiety and depression status. The Hospital Anxiety and Depression (HAD) scale will be used to assess Anxiety and Depression, which is a well-documented tool for assessing symptoms of anxiety and depression in patients with somatic diseases.

DETAILED DESCRIPTION:
AIM (S) / OBJECTIVE OF STUDY

1. To compare the prevalence of anxiety and depression in patients with sleep disorders (OSA), COPD and the general population of North West Adelaide.
2. To study the effect of CPAP on depression and anxiety in patients with sleep apnoea who also have anxiety and depression.

STUDY DESIGN/ SETTING/LOCATION/POPULATION

This is a multicenter Prospective Cohort study run at the Lyell McEwin Hospital (LMH) and The Queen Elizabeth Hospital (TQEH), among patients attending the Respiratory and Sleep Outpatient Clinics at the Lyell McEwin Hospital (LMH) and The Queen Elizabeth Hospital (TQEH). These both sites are teaching tertiary hospital.

STUDY OUTCOMES

1. Primary Outcome To establish the prevalence of anxiety and depression in patients with sleep disorders and compare how this prevalence differs from its prevalence in COPD and in the general population.
2. Secondary Outcome To evaluate whether treatment with CPAP improves anxiety and depression symptoms (HAD scale) at 3 and 12 months in OSA patients with anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Respiratory and Sleep Outpatient Clinics at LMH and TQEH with OSA or COPD
* Aged over 18 years

Exclusion Criteria:

* Unwilling or unable to give informed written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
To establish the prevalence of anxiety and depression in patients with sleep disorders and compare how this prevalence differs from its prevalence in COPD and in the general population. | 24weeks

SECONDARY OUTCOMES:
To evaluate whether treatment with CPAP improves anxiety and depression symptoms (HAD scale) at 3 and 12 months in OSA patients with anxiety and depression. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Ameer, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- The Queen Elizabeth Hospital, Adelaide, South Australia, Australia